CLINICAL TRIAL: NCT03253874
Title: Evaluation of a Choosing Wisely™ Intervention to Reduce Low Value Pre-Operative Care for Patients Undergoing Cataract Surgery
Brief Title: Pre-Operative Testing for Cataract Surgery Among Adults in LA County
Acronym: CW-CATARACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government); LAC+USC Medical Center (Other)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UCLA IRB #16-000932
Record Dates: First submitted 2016-11-15; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Cataract
Keywords: Pre-operative Testing; Cataract Surgery; Health Service Research; Low-Value Care; Safety-Net Hospital
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Site-LAC+USC Medical Center (Experimental): In this arm or study site,new guidelines are disseminated to all residents attending and faculty physicians within the department of Ophthalmology and Anesthesiology. New guidelines call for the across the board elimination of pre-operative testing and visits for patients undergoing cataract surgery.
  Interventions: Behavioral: No Pre-Op Testing for Cataract Surgeries
- Control Site--Harbor-UCLA Medical Center (No Intervention): In this arm or study site, patients will undergo standard of care for cataract surgery without any new guidelines.

INTERVENTIONS:
Behavioral: No Pre-Op Testing for Cataract Surgeries — Supported by the American Board of Internal Medicine's Choosing Wisely™ campaign to reduce low value care , the interventions aims to reduce pre-operative visits and testing for patients undergoing cataract surgeries.
  Arms: Intervention Site-LAC+USC Medical Center

SUMMARY:
A multi-disciplinary intervention will reduce inappropriate preoperative testing for cataract surgery. Despite multiple rigorous randomized controlled trials and meta-analyses showing that pre-operative testing for cataract surgery does not improve outcomes, pre-operative testing has not declined. A quality improvement initiative, which includes gaining senior leadership support, changing the culture of care, and elimination of pre-operative consultation visits for cataract surgery, to reduce inappropriate pre-operative testing. Quasi-experimental difference-in-difference analysis comparing the intervention arm (LAC+USC Medical Center) with the control arm (Harbor-UCLA Medical Center), 6 months prior and 6 months after the intervention. Generalized estimating equation models will adjust for age, gender, race/ethnicity, comorbidities and cluster by site.

DETAILED DESCRIPTION:
Pre-operative testing for cataract surgery provides no discernible benefit to patients, increases risk of harm, and substantially raises healthcare costs-representing the quintessential example of low value care. Despite multiple randomized controlled trials demonstrating no benefit, physicians continue to routinely order pre-operative testing for most patients undergoing cataract surgery.

Supported by the American Board of Internal Medicine's Choosing Wisely™ campaign to reduce low value care, a quality improvement (QI) initiative to reduce pre-operative visits and testing for cataract surgery at LAC+USC Medical Center, a safety-net health system serving Los Angeles County's under-resourced populations and control site, Harbor-UCLA Medical Center will be evaluated.

Using Institute for Healthcare Improvement PDSA (plan, do, study, act) cycle techniques, the QI team implemented the following steps (1) review randomly sampled charts on cataract surgery patients, (2) show local data on over-testing to hospital leadership, (3) obtain buy-in from the chairs of anesthesia and ophthalmology, (4) recruit an ophthalmology resident champion, and (5) empower nurses to stop scheduling pre-operative visits for cataract surgery. On October 13th, 2015, at LAC+USC Medical Center but not Harbor-UCLA, the resident champion and department chairs emailed "new" clinical guidelines for pre-operative testing to faculty, trainees, and staff, and specifically promoted avoidance of pre-operative testing for cataract surgery, except for guideline-concordant point-of-care glucose testing for patients with diabetes and potassium testing for patients with chronic kidney disease.

Evaluation of this quality improvement initiative will consists of a quasi-experimental pre-post time series analysis. Primary outcomes include pre-operative medical visits, laboratory testing, chest X-rays and electrocardiograms within 80 days of surgery (chart review revealed the maximum duration of pre-operative testing was 80 days) for patients undergoing cataract surgery before and after the intervention.

Multivariable generalized linear models that account for clustering by clinician and adjust for patient and provider characteristics and time (in months) will be used.

.

ELIGIBILITY:
Inclusion Criteria:

* Any DHS patient scheduled for cataract surgery over the 24 month time period

Exclusion Criteria:

* DHS patient who are not undergoing cataract surgery over the last 24 months period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1798 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Inappropriate pre-operative testing (Clinical Labs) | 1 year: 6 months prior to guideline implantation & 6 month after guideline implementation
  Electronic health records will be used to identify patients with a CPT (procedure) code for cataract surgery. Using CPT (procedure) codes for pre-preoperative clinical laboratory tests (Comprehensive Metabolic Panel, CBC Plate Diff). Using CPT (procedure) codes for pre-preoperative EKGs procedures. Using CPT (procedure) codes for pre-preoperative Chest X-rays. Using CPT (procedure) codes for pre-preoperative Provider Visits (LVN/RN/PA) Visits.
Inappropriate pre-operative testing (EKG) | 1 year: 6 months prior to guideline implantation & 6 month after guideline implementation
  Electronic health records will be used to identify patients with a CPT (procedure) code for cataract surgery. Using CPT (procedure) codes for pre-preoperative EKGs procedures.
Inappropriate pre-operative testing (Chest X-rays) | 1 year: 6 months prior to guideline implantation & 6 month after guideline implementation
  Electronic health records will be used to identify patients with a CPT (procedure) code for cataract surgery. Using CPT (procedure) codes for pre-preoperative Chest X-rays.
Inappropriate pre-operative testing (Provider Visits) | 1 year: 6 months prior to guideline implantation & 6 month after guideline implementation
  Electronic health records will be used to identify patients with a CPT (procedure) code for cataract surgery. Using CPT (procedure) codes for pre-preoperative Provider Visits (LVN/RN/PA) Visits.

SECONDARY OUTCOMES:
Adverse post-operative events (e.g., arrhythmia, hyperkalemia, etc). | 1 year: 6 months prior to guideline implantation & 6 month after guideline implementation
  Complications or adverse event s during surgery, and after surgery (30 day). New ICD Diagnostic codes will be explore 30 days after surgery or date of surgery to determine if there are any adverse events/surgical complications. Adverse events post-operative will be monitored to ensure the intervention is not leading to harm.
Time to Surgery | 1 year: 6 months prior to guideline implantation & 6 month after guideline implementation
  Wait-times starting from diagnosis of cataracts until surgery

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A. Sarkisian, MD, MSHS, Principal Investigator — University of California, Los Angeles